CLINICAL TRIAL: NCT00026494
Title: A Phase I/II Trial Of Temozolomide And Vinorelbine For Patients With Recurrent Brain Metastases
Brief Title: Temozolomide and Vinorelbine in Treating Patients With Recurrent Brain Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-088; MSKCC-01088A; NCI-G01-2025
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Temozolomide; Vinorelbine

ARMS (1):
- Temozolomide and Vinorelbine (Experimental): Patients will be treated with vinorelbine on days 1 and 8 of each cycle; temozolomide will be administered on days 1 to 7 and 15 to 21 of each cycle. The dose level of temozolomide will be given at a dose of 150 mg/m2/day. A cycle will be defined as 28 days of treatment.
  Interventions: Drug: temozolomide; Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: temozolomide
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of temozolomide and vinorelbine in treating patients who have recurrent brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of vinorelbine when administered in combination with temozolomide in patients with recurrent brain metastases (phase I accrual completed).
* Determine the safety and feasibility of this treatment regimen in these patients.
* Determine the efficacy of this treatment regimen, in terms of objective radiographic response and overall and progression-free survival, in these patients.

OUTLINE: This is a dose-escalation study of vinorelbine.

Patients receive vinorelbine IV over 5-10 minutes on days 1 and 8 and oral temozolomide once daily on days 1-7 and 15-21. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of vinorelbine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 20-35 patients will be treated at that dose level.

Patients are followed every 3-4 months.

PROJECTED ACCRUAL: A minimum of 3 patients will be accrued for the phase I portion of this study and 20-35 patients will be accrued for the phase II portion of this study within 2 years.

ELIGIBILITY:
INCLUSION CRITERIAL:

* Age > or = 18 years.
* Karnofsky performance score > or = 60.
* Histopathologic confirmation of the diagnosis of a solid tumor malignancy. The brain metastasis diagnosis per se does not have to be pathologically confirmed if the clinical and neuro radiographic picture is typical.
* MRI (or CT if the patient cannot undergo MRI) evidence of evaluable disease in the brain.
* Absolute neutrophil count > or = 1,500/mm³. Platelet count > or = 100,000/mm³.
* Hemoglobin > or = 10 g/dl.
* BUN and serum creatinine both < 1.5 times upper limit of normal.
* Total and direct bilirubin both < 1.5 times upper limit of normal.
* SGOT and SGPT both < or = 3 times upper limit of normal.
* Alkaline phosphatase < or = 2 times upper limit of normal.
* At least two weeks must have elapsed from brain biopsy, craniotomy, or other surgery.
* Life expectancy > or = 8 weeks.
* Patient or their legal guardian or legal next-of-kin must provide written informed consent prior to patient's registration on study.
* At least four weeks must have elapsed from previous external beam radiation therapy, or eight weeks from stereotactic radiosurgery.
* Patients treated with radiosurgery should have evidence of progression at a distant site in the brain, or confirmation of tumor progression by biopsy or PET scan.

EXCLUSION CRITERIA:

* Previous treatment with temozolomide, dacarbazine or vinorelbine.
* Patients who have not recovered from all acute toxicities of prior therapies.
* Patients with evidence of leptomeningeal metastases or primary dural metastases.
* Patients who are poor medical risks because of nonmalignant systemic disease, as well as those with acute infection requiring treatment with intravenous antibiotics.
* Patients whose psychiatric condition would, in the judgment of the principal investigator, make it unlikely that they could adhere to the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2001-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E. Abrey, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Iwamoto FM, Omuro AM, Raizer JJ, Nolan CP, Hormigo A, Lassman AB, Gavrilovic IT, Abrey LE. A phase II trial of vinorelbine and intensive temozolomide for patients with recurrent or progressive brain metastases. J Neurooncol. 2008 Mar;87(1):85-90. doi: 10.1007/s11060-007-9491-3. Epub 2007 Nov 7. PMID 17987262

RESULTS

PARTICIPANT FLOW:
Groups:
- 15mg/m2 - Vinorelbine: Temozolomide and 15mg/m2 Vinorelbine for Patients with Recurrent Brain Metastases
- 20mg/m2 - Vinorelbine: Temozolomide and 20mg/m2 Vinorelbine for Patients with Recurrent Brain Metastases
- 25mg/m2 - Vinorelbine: Temozolomide and 25mg/m2 Vinorelbine for Patients with Recurrent Brain Metastases
- 30mg/m2 - Vinorelbine: Temozolomide and 30mg/m2 Vinorelbine for Patients with Recurrent Brain Metastases
Period: Overall Study
Arm/Group | 15mg/m2 - Vinorelbine | 20mg/m2 - Vinorelbine | 25mg/m2 - Vinorelbine | 30mg/m2 - Vinorelbine
Started | 7 | 4 | 22 | 16
Completed | 5 | 4 | 16 | 16
Not Completed | 2 | 0 | 6 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Patient non-compliance | 1 | 0 | 0 | 0
Not completed — Patient not treated | 0 | 0 | 2 | 0
Not completed — Clinical progression | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15mg/m2 - Vinorelbine | 20mg/m2 - Vinorelbine | 25mg/m2 - Vinorelbine | 30mg/m2 - Vinorelbine | Total
Number analyzed (Participants) | 7 | 4 | 22 | 16 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 17 | 10 | 34
  >=65 years | 2 | 2 | 5 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 13 | 10 | 29
  Male | 2 | 3 | 9 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Assessed by Macdonald Criteria Every 2 Months
Description: All patients will have their tumor measurements recorded at baseline and at the time of each MRI scan. Lesions must be measured in two dimensions.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | 15mg/m2 - Vinorelbine | 20mg/m2 - Vinorelbine | 25mg/m2 - Vinorelbine | 30mg/m2 - Vinorelbine
Number analyzed (Participants) | 5 | 4 | 16 | 16
participants
  Stable Disease (SD) | 3 | 2 | 4 | 3
  Progression of Disease (POD) | 2 | 1 | 11 | 12
  Partial Response (PR) | 0 | 1 | 0 | 0
  Minor Response (MR) | 0 | 0 | 1 | 0
  Complete Response (CR) | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | 15mg/m2 - Vinorelbine | 20mg/m2 - Vinorelbine | 25mg/m2 - Vinorelbine | 30mg/m2 - Vinorelbine
Serious Adverse Events (participants affected / at risk) | 4/7 | 4/4 | 8/22 | 9/16
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 19/22 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15mg/m2 - Vinorelbine (N=7) | 20mg/m2 - Vinorelbine (N=4) | 25mg/m2 - Vinorelbine (N=22) | 30mg/m2 - Vinorelbine (N=16)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1) | 4 (7)
Supravent arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Leukocytes (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 4 (7)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Syncope (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anorexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood alteration-depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurology, other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuropathy-motor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Speech Impair (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CNS hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constitut symptoms, other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syndromes, other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15mg/m2 - Vinorelbine (N=7) | 20mg/m2 - Vinorelbine (N=4) | 25mg/m2 - Vinorelbine (N=22) | 30mg/m2 - Vinorelbine (N=16)
Abdominal pain/cramping (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Anorexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bicarbonate (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood,Bone marrow,other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CNS hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatology, skin other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hearing, other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 9 (9) | 9 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 11 (11) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesmia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 5 (5) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 5 (5)
Incontinence (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infection without neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 12 (12) | 13 (13)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 11 (11) | 12 (12)
Mood alteration-depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurology, other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neuropathy-motor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 9 (9) | 11 (11)
Ocular-Vision other (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain, other (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pelvic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Rash, desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
SGOT (AST) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
SGPT (ALT) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (5) | 6 (6)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes